CLINICAL TRIAL: NCT01909557
Title: Effect of Supplementation of Antioxidant Substances and Probiotics in HCV Correlated Liver Disease Treated With Interferon and Ribavirin. Studies on Biochemical and Virological Response and on Quality of Life.
Brief Title: Acetyl-L-Carnitine Supplementation During HCV Therapy With Peg IFN-α2b Plus Ribavirin: Effect on Work Performance.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Mariano Malaguarnera, Associate Professor, University of Catania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Unict10/1997
Record Dates: First submitted 2013-07-24; First posted 2013-07-26 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2013-07

CONDITIONS: Quality of Life; Daily Activity; Fatigue
Keywords: Acetyl-L-carnitine; Interferons; Ribavirin; Hepatitis C; Fatigue
MeSH Terms: conditions — Fatigue; Hepatitis C | interventions — Acetylcarnitine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acetyl-L-carnitine (Active Comparator): Acetyl-L-carnitine 2 gr tablets
  Interventions: Drug: Acetyl-L-carnitine
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Acetyl-L-carnitine
  Arms: Acetyl-L-carnitine
Drug: placebo
  Arms: placebo

SUMMARY:
To assess the effects of Acetyl-L-Carnitine, probiotics and antioxidant nutritional substances administration on work productivity, daily activity, and fatigue in subjects with chronic hepatitis C treated with Pegylated-Interferon-α2b and Ribavirin.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients are workers who are 18 years of age or older, infected by HCV with a quantifiable serum HCV RNA level (as determined by polimerase chain reaction, COBAS AmpliPrep/COBAS TaqMan - ROCHE). HCV infected populations must have elevated serum alanine transaminase levels and findings on liver biopsy consistent with chronic infection. Cirrhotic patients have to have a Child-Pugh score less than 7 to be eligible.

Exclusion Criteria:

* Ineligible patients are those who had other liver diseases, as well as those who are affected by cancer, severe jaundice, pulmonary and renal chronic diseases, prostatic diseases, autoimmune diseases and diabetes mellitus. Excessive use of alcohol (>20 g/die) or hepato-toxic drugs. Other causes of exclusion include decompensated cirrhosis, pregnancy, and contraindications for Peg-IFN-a or RBV therapy such as cardiopathy, hemoglobinopathies, hemocromatosis, major depression or other severe psychiatric pathological conditions.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Work performances | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Catania, Cannizzaro Hospital, Catania, Italy